CLINICAL TRIAL: NCT05161039
Title: Recoil Feasibility Study for the Treatment of Atherosclerotic Lesions in the Infrapopliteal Arteries Comparing Serration Angioplasty (Serranator® Device) vs. Plain Balloon Angioplasty (POBA)
Brief Title: Serranator Recoil Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cagent Vascular LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CSP-0485
Record Dates: First submitted 2021-11-19; First posted 2021-12-16 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Peripheral Arterial Disease; Critical Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Serranator (Other)
  Interventions: Device: Serranator
- POBA (Other)
  Interventions: Device: POBA

INTERVENTIONS:
Device: Serranator — Serranator® PTA Serration Balloon Catheter manufactured by Cagent Vascular
  Arms: Serranator
Device: POBA — Plain balloon angioplasty device
  Arms: POBA

SUMMARY:
The study objective is to assess the ability to define and measure post treatment recoil in infrapopliteal arteries. Preliminary evidence as to the differences between serration angioplasty and standard balloon angioplasty as defined by post treatment recoil, lumen gain, and dissection will be collected.

DETAILED DESCRIPTION:
Multi-center, feasibility study treating up to 20 atherosclerotic lesions in the infrapopliteal arteries. The study will capture angiographic imaging (pre, during, post, and post 15 mins) for all lesions, and a subset (up to 10) of IVUS imaging data (pre, post, and post 15 mins), to compare serration angioplasty vs standard angioplasty and its effects on vessel recoil and final diameter stenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of >18 years old.
2. Women of childbearing potential must have a negative urine pregnancy test within 7 days of index procedure.
3. Subject or subject's legal representative has been informed of the nature of the study, agrees to participate, and comply, and has signed the consent form.
4. Subject has Rutherford Clinical Category 3, 4, 5, or 6.

Angiographic Inclusion Criteria:

1. Target lesion(s) has stenosis >70% by visual assessment;
2. De-novo, or non-stented re-stenotic lesions;
3. Reference vessel diameter is between 2.5 mm and 3.5 mm, inclusive;
4. Target lesions involve infrapopliteal tibial arteries including pedal;
5. A target lesion may consist of one long or multiple serial lesions that are up to and including 12 cm in length;
6. If a second lesion is identified in another vessel, the second lesion can also be treated and if treated will be treated with the alternate treatment.

Exclusion Criteria:

1. Evidence of aneurysm or acute thrombus in the target vessel.
2. Subject has an allergy to contrast medium that cannot be pretreated.
3. Subject is pregnant or breastfeeding.

Angiographic Exclusion Criteria:

1. Acute Total Occlusions; evidence of acute thrombus formation by angiography.
2. In-stent restenotic lesions.
3. Inability to cross the lesion with the assigned study device.
4. Treatment of target lesion with atherectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Presence of post treatment recoil | 15 minutes post procedure
  Obtain preliminary data on post treatment recoil in infrapopliteal arteries utilizing angiographic and IVUS data following serration angioplasty and standard angioplasty.

CONTACTS AND LOCATIONS:
Locations (2):
- Stanford University, Palo Alto, California, United States
- Klinik für Angiologie, Klinikum Hochsauerland GmbH, Arnsberg, Germany